CLINICAL TRIAL: NCT06839144
Title: Inhibiting Beta-adrenergic and COX-2 Signaling During the Perioperative Period to Reduce Ovarian Cancer Progression: A Randomized Placebo-Controlled Clinical Trial
Brief Title: Inhibiting Beta-adrenergic and COX-2 Signaling During the Perioperative Period to Reduce Ovarian Cancer Progression
Acronym: OC-POP-PT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: National Cancer Institute (NCI) (NIH); The Chaim Sheba Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLV-0199-24; 1R21CA291683-01 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; Ovarian Cancer Metastatic Recurrent
Keywords: Ovarian Cancer; Perioperative Intervention; Beta-Blockers; Propranolol; COX-2 Inhibitors; Etodolac; Psychoneuroimmunology; Stress and Cancer; Randomized Controlled Trial (RCT); Biomarker Analysis
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Propranolol; Adrenergic beta-Antagonists; Etodolac; Cyclooxygenase 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Patients receive propranolol + etodolac (active treatment)
  Interventions: Drug: Propranolol (Beta-Blocker) and Etodolac (COX-2 Inhibitor)
- Placebo Arm (Placebo Comparator): Patients receive matching placebo for both drugs
  Interventions: Drug: Placebo (Matching for Propranolol & Etodolac)

INTERVENTIONS:
Drug: Propranolol (Beta-Blocker) and Etodolac (COX-2 Inhibitor) — - Intervention Arm: Propranolol (Beta-Blocker) and Etodolac (COX-2 Inhibitor). Name: Propranolol (slow-Release) and Etodolac.
  Propranolol Dosage Schedule:
  5 days pre-surgery: 20mg twice daily (BID), Day of surgery: 80mg BID,
  1-week Post-surgery: 40mg BID, week 2-11 post-surgery: 20mg BID.
  Etodolac Dosage Schedule:
  5 days pre-surgery until 3 weeks post-surgery: 400mg BID.
  Administration Route: Oral.
  Arms: Intervention Arm
Drug: Placebo (Matching for Propranolol & Etodolac) — - Placebo Arm: Placebo (Matching for Propranolol & Etodolac). Inert placebo tablets matching propranolol and etodolac in appearance and dosing schedule. Administration Route: Oral.
  Arms: Placebo Arm

SUMMARY:
This study investigates the impact of perioperative inhibition of beta-adrenergic and COX-2 signaling in ovarian cancer patients undergoing debulking surgery. The trial aims to assess the feasibility, safety, and biological effects of a combination of propranolol and etodolac in reducing cancer metastasis and improving immune responses.

DETAILED DESCRIPTION:
The study is a placebo-controlled randomized clinical trial (RCT) enrolling 60 women undergoing ovarian cancer debulking surgery. Participants will be assigned to receive propranolol (starting 5 days preoperatively, increased on the day of surgery, and continued postoperatively) and etodolac at a fixed dose. The primary outcomes include recruitment rate, drug safety, tolerability, adherence, and molecular tumor and blood characteristics. Secondary outcomes include 3-year recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-85
* ASA score 1-3 or ECOG Performance Status of 0 to 2
* Patients with a suspected high-grade ovarian epithelial cancer based on imaging, clinical examination, CA125, and/or tumor biopsy
* Patients planned for surgery for primary surgery, or interval debulking surgery for ovarian cancer
* Signed informed consent form
* Willing and able to comply with study procedures (physically and mentally)

Exclusion Criteria:

* Patients who participate in another interventional study
* Patients with known allergy to one or more of the study medications, or to any medication from the non-steroidal anti-inflammatory drug group or beta-blockers family
* Patients treated chronically with any type of a beta-adrenergic blocker or a COX inhibitor, except use of Aspirin, which will be discontinued at least 7 days prior to surgery, and until 3 weeks post-surgery
* Patients currently suffering from asthma (אסתמה פעילה בלבד), or required hospital admission or change in medical treatment for asthma within the past year
* Patients with active peptic disease
* Patients with a history of CVA/TIA
* Recent (within the last 5 years) or concurrent malignancies, with the exception of adequately treated in-situ carcinoma of the cervix or basal-cell carcinoma of the skin
* Patients with renal failure, measured by creatinine level >1.5
* Patients with significant liver dysfunction (known cirrhosis, Bilirubin level>2)
* Patients with significant heart failure (NYHA functional class 3 or Higher)
* Patients with bradycardia (heart rate of 50 or less) or second- or third-degree AV block
* Patients with right-sided heart failure owing to pulmonary hypertension
* Patients with chronic Digoxin treatment
* Patients with Printzmetal's angina
* Patients with significant diagnosed cardiomegaly
* Patients suffering from sick sinus syndrome
* Patients with peripheral vascular disease
* Patients with current (unresected) pheochromocytoma
* Pregnant women
* Patients who are treated with immunosuppressive medications, including chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial drug
* Patients with Immunodeficiency Disorders

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Transcriptional Activity in Excised Tumors | At the time of surgery (Day 0). Data will be reported through study completion, an average of 2 years.
  Transcriptional activity related to pro-metastatic (e.g., EMT), pro-growth (STAT and GATA families), and stress and inflammatory signaling (NF-κB/cRel, AP-1, CREB, GR) in excised tumors.
Transcriptional Activity in Blood Samples | Preoperative baseline (Informed consent day), Day 0 (surgery), postoperative Day 1, Week 3, and Week 11. Data will be reported through study completion, an average of 2 years.
  Longitudinal analysis of transcriptional activity in peripheral blood, focusing on stress/inflammatory pathways (NF-κB/cRel, AP-1, CREB, GR). Unit of measure: Relative expression levels (fold change).
Adverse Event Assessment | From 5 days pre-surgery to 3 months post-surgery.
  Recording and categorization of adverse events, using a standardized tool (e.g., CTCAE-Common Terminology Criteria for Adverse Events) to assess the severity and type of adverse events. Unit of Measure: Number and severity of adverse events.
Patient Adherence to Drug Regimen | From 5 days pre-surgery to 3 months post-surgery.
  Patient adherence will be assessed using pill counts or patient self-reports. Unit of Measure: Percentage of prescribed dosage consumed.
Recruitment Rate | Study duration (estimated 2 years).
  Number of participants enrolled in the study within the specified timeframe.

SECONDARY OUTCOMES:
Three-Year Recurrence Rate | 3 years post-surgery.
  Assessment of recurrence in patients based on medical records and follow-ups at 3 years post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nadav Michaan, Prof., Principal Investigator — Tel Aviv Sourasky Medical Center (Ichilov Hospital); Anna Blecher, Dr., Principal Investigator — The Chaim Sheba Medical Center (Tel Hashomer); Shamgar Ben-Eliyahu, Prof., Principal Investigator — Tel Aviv University
Locations (2):
- Israel (2):
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center (Ichilov Hospital), Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: Within 12 months of study completion and final data analysis.
Access Criteria: Upon request via data-sharing agreements through Tel Aviv University.

REFERENCES:
- [Background] Shaashua L, Shabat-Simon M, Haldar R, Matzner P, Zmora O, Shabtai M, Sharon E, Allweis T, Barshack I, Hayman L, Arevalo J, Ma J, Horowitz M, Cole S, Ben-Eliyahu S. Perioperative COX-2 and beta-Adrenergic Blockade Improves Metastatic Biomarkers in Breast Cancer Patients in a Phase-II Randomized Trial. Clin Cancer Res. 2017 Aug 15;23(16):4651-4661. doi: 10.1158/1078-0432.CCR-17-0152. Epub 2017 May 10. PMID 28490464
- [Background] Haldar R, Ricon-Becker I, Radin A, Gutman M, Cole SW, Zmora O, Ben-Eliyahu S. Perioperative COX2 and beta-adrenergic blockade improves biomarkers of tumor metastasis, immunity, and inflammation in colorectal cancer: A randomized controlled trial. Cancer. 2020 Sep 1;126(17):3991-4001. doi: 10.1002/cncr.32950. Epub 2020 Jun 13. PMID 32533792
- [Background] Haldar R, Shaashua L, Lavon H, Lyons YA, Zmora O, Sharon E, Birnbaum Y, Allweis T, Sood AK, Barshack I, Cole S, Ben-Eliyahu S. Perioperative inhibition of beta-adrenergic and COX2 signaling in a clinical trial in breast cancer patients improves tumor Ki-67 expression, serum cytokine levels, and PBMCs transcriptome. Brain Behav Immun. 2018 Oct;73:294-309. doi: 10.1016/j.bbi.2018.05.014. Epub 2018 May 22. PMID 29800703